CLINICAL TRIAL: NCT01668758
Title: Detection of Hemodynamic Changes in Traumatic Brain Injuries Population With Functional Near Infrared Spectroscopy
Brief Title: fMRI and NIRS Imaging for Traumatic Brain Injury
Status: Withdrawn | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120165; 12-CH-0165
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2013-07-01

CONDITIONS: Cognition Disorder; Functional Brain Imaging
Keywords: Near Infrared Spectroscopy; Traumatic Brain Injury
MeSH Terms: conditions — Cognition Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- The amount of blood flowing in brain areas goes up when those areas are being used for activities, such as movement or seeing. Functional magnetic resonance imaging (fMRI) is a common way of measuring blood flow in the brain. Near infrared spectroscopy (NIRS) can also be used to study blood flow in the brain. However, NIRS has not been used as often as fMRI. Researchers want to compare fMRI and NIRS to see whether they give similar results. These studies will be used to look at people who have had a traumatic brain injury.

Objectives:

- To test how well NIRS measure changes in blood flow in the brain after a traumatic brain injury.

Eligibility:

* Individuals between 18 and 60 years of age who have had a traumatic brain injury.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Researchers may ask to see brain images during from previous MRI scans.
* Participants will have a NIRS scan of the brain. They will be asked to do certain tasks while inside the scanner. These tasks will involve responding to images that appear on a screen.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
The goal of this study is to be able to assess frontal lobe function in a rapid, objective, and standardized way, without the need for expertise in cognitive test administration. Such methods would be particularly helpful in mild traumatic brain injury, where objective measures are needed, and would greatly expand the capacity to make such assessments in standard clinical practice.

Our goal is to recruit 100 subjects total in two groups of age, gender, and education matched subjects, as follows: TBI (n = 50) and non-TBI (n = 50).

The subject will be asked to perform 2 computer-based cognitive tests while the fNIRS device is in place. The fNIRS sensor pads will record changes in blood oxy/deoxy hemoglobin concentrations in the underlying cortex. Data will be stored for post processing analysis.

The main outcome measures will be: 1) a correlation of the fNIRS results between the TBI and non-TBI groups; 2) a correlation of the fNIRS results with the severity of the TBI within the TBI group. Finally, we plan to compare individual measurement from TBI patients with the healthy group.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy population

- Age 18 to 60, inclusive.

Traumatic brain injuries population

* Age 18 to 60.
* Have a recorded past traumatic brain injuries rated in the Glasgow Coma Scale between 9 and 15

EXCLUSION CRITERIA:

* Pregnancy
* History of hypertension
* History of any disease of the central nervous system
* Current use of sedating medication, including antihistamines
* Subjects with any of the following will be excluded from MRI testing: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or autodefibrillator; cochlear implant; ocular foreign body, such as metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing due to the possible dangerous effects of the MRI magnet upon metal objects in the body.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-25; Study Completion 2013-07-01

PRIMARY OUTCOMES:
The main outcome measures will be to identify if the brain flow hemodynamic between the healthy and the TBI group is affected by trauma.

SECONDARY OUTCOMES:
The secondary outcome of the two parametric paradigms will investigate if the degree of disruption correlates with measures of the severity of injury (GC scale). Finally, we will compare individual measurement form TBI patient with the health...

CONTACTS AND LOCATIONS:
Overall Officials: Amir Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)

REFERENCES:
- [Background] Hanna-Pladdy B. Dysexecutive syndromes in neurologic disease. J Neurol Phys Ther. 2007 Sep;31(3):119-27. doi: 10.1097/NPT.0b013e31814a63c2. PMID 18025957
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Strangman GE, Goldstein R, O'Neil-Pirozzi TM, Kelkar K, Supelana C, Burke D, Katz DI, Rauch SL, Savage CR, Glenn MB. Neurophysiological alterations during strategy-based verbal learning in traumatic brain injury. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):226-36. doi: 10.1177/1545968308324225. Epub 2008 Dec 1. PMID 19047359